CLINICAL TRIAL: NCT04673422
Title: Effect of Montelukast in Preventing Dengue With Warning Signs in Dengue Patients: a Multicenter Randomized, Double-blind, Placebo Controlled, Superiority Trial
Brief Title: Effect of Montelukast in Preventing Dengue With Warning Signs in Dengue Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Phramongkutklao College of Medicine and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AMEDDengue2020
Record Dates: First submitted 2020-12-09; First posted 2020-12-17 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Dengue; Dengue With Warning Signs; Dengue Shock Syndrome
MeSH Terms: conditions — Dengue; Severe Dengue | interventions — montelukast

STUDY DESIGN:
Intervention Model Description: a randomized, prospective, 2-arm, parallel-group, double-blind, placebo-controlled superiority trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Montelukast (Experimental): a 10 mg tablet will be given orally immediately and every day thereafter for 10 days or until recovery, defined as the discontinuation of the follow up appointment by the attending physicians, whichever is shorter
  Interventions: Drug: Montelukast
- Placebo (Placebo Comparator): a 10 mg tablet will be given orally immediately and every day thereafter for 10 days or until recovery, defined as the discontinuation of the follow up appointment by the attending physicians, whichever is shorter
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Montelukast — A 10-mg tablet will be given orally immediately and every day thereafter for 10 days or until recovery, defined as the discontinuation of the follow up appointment by the attending physicians, whichever is shorter
  Arms: Montelukast
Drug: Placebo — A 10-mg tablet will be given orally immediately and every day thereafter for 10 days or until recovery, defined as the discontinuation of the follow up appointment by the attending physicians, whichever is shorter
  Arms: Placebo

SUMMARY:
This study aims to determine the efficacy of montelukast in reducing the incidence of dengue warning signs in adult dengue patients.

DETAILED DESCRIPTION:
Dengue has been the growing public health problem in many tropical countries. Almost 4 billion people were estimated to be at risk, with estimated 400 million infections occurring annually. In Asia, around 10% of febrile patients were virologically confirmed with dengue. The most common cause of death is from dengue shock as a result of vascular leak syndrome. This condition can occur in various clinical manifestations ranging from mild cases to life-threatening condition of dengue shock syndrome. The common sites of plasma leakage are pleural effusion and ascites. The contributing factors for endothelial dysfunction in dengue are cytokines such as soluble tumor necrosis factor receptor (sTNFR/75), interferon gamma, and vascular endothelial growth factor, NS1 antigenemia, complement activation, and activation of dendritic cells, macrophages, and mast cells.

Mast cells have recently been acknowledged as an important regulator for promoting innate immune responses. Important composition of granules in mast cells are proteases, chymase and tryptase, histamine, heparin and leukotriene. The activated mast cells can undergo degranulation, releasing these cytokines. These increase capillary permeability, leading to vascular leakage.

Leukotriene has an important role in promoting plasma leakage and leukocyte adhesion in postcapillary venules. In dengue patients, leukotriene levels usually elevate during febrile and defervescence stage for 35 and 38 times of the baseline values, and return to baseline in convalescence stage. Blocking leukotriene in dengue infected mice can significantly reduce plasma leakage.

The management of dengue consists of only symptomatic treatment, and intravenous fluid replacement. No specific treatment has yet been demonstrated of a benefit in preventing complications. In the recent decades, mast cells have been demonstrated as a major contributor of severe forms of dengue, leading to research in reduction of vascular permeability with mast cell stabilizers or anti-histamine drugs. An animal model studies found that a tryptase inhibitor, nafamostat, or leukotriene inhibitor, montelukast, could reduce the plasma leakage.

In 2018, an open-label study found that patients with montelukast had a 22% absolute risk reduction in dengue shock syndrome, compared to standard treatment. However, there has never been any randomized controlled trial evaluating the efficacy of montelukast in dengue patients.

This study aims to determine the efficacy of montelukast in reducing the incidence of dengue warning signs in adult dengue patients.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* diagnosis of dengue
* positive NS1 antigen or polymerase chain reaction (PCR) test

Exclusion Criteria:

* any warning sign of dengue
* concurrent diagnosis of other causes of fever, such as malaria or heat stroke
* pregnancy
* being unable to take medication by mouth
* critical illness needing intubation or admission to an intensive care unit
* being unable to communicate
* other indication of montelukast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2023-06-17 (Actual); Study Completion 2023-06-17 (Actual)

PRIMARY OUTCOMES:
Rate of dengue with warning signs | 14 days or until the discontinuation of the follow up appointment by the attending physicians, whichever is shorter.
  Rate of a composite outcome including
  * abdominal tenderness or pain
  * persistent vomiting
  * clinical fluid accumulation
  * mucosal bleeding
  * liver enlargement >2cm
  * increase in hematocrit concurrent with decrease in platelet count However, lethargy will be excluded as a criterion for warning sign as almost all patients reported subjective lethargy.

SECONDARY OUTCOMES:
Rate of each component of composite outcome of dengue with warning signs | 14 days or until the discontinuation of the follow up appointment by the attending physicians, whichever is shorter
  Rate of each component of composite outcome of dengue with warning signs
  * abdominal tenderness or pain
  * persistent vomiting
  * clinical fluid accumulation
  * mucosal bleeding
  * liver enlargement >2cm
  * increase in hematocrit concurrent with decrease in platelet count
Rate of hospitalization | 14 days or until the discontinuation of the follow up appointment by the attending physicians, whichever is shorter
  Rate of admission to hospital
Length of hospital stay | up to 90 days
  Length of hospital stay
Rate of severe dengue | 14 days or until the discontinuation of the follow up appointment by the attending physicians, whichever is shorter
  Rate of a composite outcome including
  * shock
  * fluid accumulation with respiratory distress
  * severe bleeding leading to hypotension or decreased hematocrit
  * liver transaminase >1000
  * impaired consciousness
  * heart and other organ failure
Rate of dengue shock | 14 days or until the discontinuation of the follow up appointment by the attending physicians, whichever is shorter
  Rate of hypotension or the pulse pressure of ≤ 20 mm Hg
30-day mortality | 30 days
  death with in 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Worapong Nasomsong, MD, Principal Investigator — Phramongkutklao College of Medicine and Hospital; Worayon Chuerboonchai, MD, Principal Investigator — Ananda Mahidol Hospital
Locations (4):
- Thailand (4):
  - Hatyai Hospital, Hat Yai, Changwat Songkhla
  - Phramongkutklao Hospital, Bangkok
  - Ananda Mahidol Hospital, Lopburi
  - Fort Suranari Hospital, Nakhon Ratchasima

IPD SHARING:
Plan to Share IPD: Yes
Data requests can be made anytime from 6 months after the publication of this trial. De-identified participant data can be requested by researchers for use in independent scientific research and will be provided following review and approval of the research proposal (including statistical analysis plan).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: starting 6 months after publication
Access Criteria: De-identified participant data can be requested by researchers for use in independent scientific research and will be provided following review and approval of the research proposal (including statistical analysis plan). Requests should be sent to the corresponding author after publication.

REFERENCES:
- [Background] Guzman MG, Gubler DJ, Izquierdo A, Martinez E, Halstead SB. Dengue infection. Nat Rev Dis Primers. 2016 Aug 18;2:16055. doi: 10.1038/nrdp.2016.55. PMID 27534439
- [Background] L'Azou M, Moureau A, Sarti E, Nealon J, Zambrano B, Wartel TA, Villar L, Capeding MR, Ochiai RL; CYD14 Primary Study Group; CYD15 Primary Study Group. Symptomatic Dengue in Children in 10 Asian and Latin American Countries. N Engl J Med. 2016 Mar 24;374(12):1155-66. doi: 10.1056/NEJMoa1503877. PMID 27007959
- [Background] Wilder-Smith A, Ooi EE, Horstick O, Wills B. Dengue. Lancet. 2019 Jan 26;393(10169):350-363. doi: 10.1016/S0140-6736(18)32560-1. PMID 30696575
- [Background] Srikiatkhachorn A, Krautrachue A, Ratanaprakarn W, Wongtapradit L, Nithipanya N, Kalayanarooj S, Nisalak A, Thomas SJ, Gibbons RV, Mammen MP Jr, Libraty DH, Ennis FA, Rothman AL, Green S. Natural history of plasma leakage in dengue hemorrhagic fever: a serial ultrasonographic study. Pediatr Infect Dis J. 2007 Apr;26(4):283-90; discussion 291-2. doi: 10.1097/01.inf.0000258612.26743.10. PMID 17414388
- [Background] Bethell DB, Flobbe K, Cao XT, Day NP, Pham TP, Buurman WA, Cardosa MJ, White NJ, Kwiatkowski D. Pathophysiologic and prognostic role of cytokines in dengue hemorrhagic fever. J Infect Dis. 1998 Mar;177(3):778-82. doi: 10.1086/517807. PMID 9498463
- [Background] Srikiatkhachorn A, Green S. Markers of dengue disease severity. Curr Top Microbiol Immunol. 2010;338:67-82. doi: 10.1007/978-3-642-02215-9_6. PMID 19802579
- [Background] Green S, Vaughn DW, Kalayanarooj S, Nimmannitya S, Suntayakorn S, Nisalak A, Lew R, Innis BL, Kurane I, Rothman AL, Ennis FA. Early immune activation in acute dengue illness is related to development of plasma leakage and disease severity. J Infect Dis. 1999 Apr;179(4):755-62. doi: 10.1086/314680. PMID 10068569
- [Background] Avirutnan P, Punyadee N, Noisakran S, Komoltri C, Thiemmeca S, Auethavornanan K, Jairungsri A, Kanlaya R, Tangthawornchaikul N, Puttikhunt C, Pattanakitsakul SN, Yenchitsomanus PT, Mongkolsapaya J, Kasinrerk W, Sittisombut N, Husmann M, Blettner M, Vasanawathana S, Bhakdi S, Malasit P. Vascular leakage in severe dengue virus infections: a potential role for the nonstructural viral protein NS1 and complement. J Infect Dis. 2006 Apr 15;193(8):1078-88. doi: 10.1086/500949. Epub 2006 Mar 9. PMID 16544248
- [Background] Nascimento EJ, Silva AM, Cordeiro MT, Brito CA, Gil LH, Braga-Neto U, Marques ET. Alternative complement pathway deregulation is correlated with dengue severity. PLoS One. 2009 Aug 26;4(8):e6782. doi: 10.1371/journal.pone.0006782. PMID 19707565
- [Background] Londono-Renteria B, Marinez-Angarita JC, Troupin A, Colpitts TM. Role of Mast Cells in Dengue Virus Pathogenesis. DNA Cell Biol. 2017 Jun;36(6):423-427. doi: 10.1089/dna.2017.3765. Epub 2017 May 9. PMID 28486041
- [Background] St John AL, Rathore AP, Yap H, Ng ML, Metcalfe DD, Vasudevan SG, Abraham SN. Immune surveillance by mast cells during dengue infection promotes natural killer (NK) and NKT-cell recruitment and viral clearance. Proc Natl Acad Sci U S A. 2011 May 31;108(22):9190-5. doi: 10.1073/pnas.1105079108. Epub 2011 May 16. PMID 21576486
- [Background] Schmutzler W, Bolsmann K, Zwadlo-Klarwasser G. Comparison of histamine release from human blood monocytes, lymphocytes, adenoidal and skin mast cells. Int Arch Allergy Immunol. 1995 May-Jun;107(1-3):194-6. doi: 10.1159/000236974. PMID 7542070
- [Background] Marone G, Varricchi G, Loffredo S, Granata F. Mast cells and basophils in inflammatory and tumor angiogenesis and lymphangiogenesis. Eur J Pharmacol. 2016 May 5;778:146-51. doi: 10.1016/j.ejphar.2015.03.088. Epub 2015 May 2. PMID 25941082
- [Background] St John AL, Rathore AP, Raghavan B, Ng ML, Abraham SN. Contributions of mast cells and vasoactive products, leukotrienes and chymase, to dengue virus-induced vascular leakage. Elife. 2013 Apr 30;2:e00481. doi: 10.7554/eLife.00481. PMID 23638300
- [Background] Syenina A, Jagaraj CJ, Aman SA, Sridharan A, St John AL. Dengue vascular leakage is augmented by mast cell degranulation mediated by immunoglobulin Fcgamma receptors. Elife. 2015 Mar 18;4:e05291. doi: 10.7554/eLife.05291. PMID 25783751
- [Background] Dahlen SE, Bjork J, Hedqvist P, Arfors KE, Hammarstrom S, Lindgren JA, Samuelsson B. Leukotrienes promote plasma leakage and leukocyte adhesion in postcapillary venules: in vivo effects with relevance to the acute inflammatory response. Proc Natl Acad Sci U S A. 1981 Jun;78(6):3887-91. doi: 10.1073/pnas.78.6.3887. PMID 6267608
- [Background] Loke WM, Chow AY, Lam Mok Sing K, Lee CY, Halliwell B, Lim EC, Quek AM, Ooi EE, Seet RC. Augmentation of 5-lipoxygenase activity and expression during dengue serotype-2 infection. Virol J. 2013 Oct 30;10:322. doi: 10.1186/1743-422X-10-322. PMID 24168271
- [Background] Sherif NA, Zayan AH, Elkady AH, Ghozy S, Ahmed AR, Omran ES, Taha EA, Eldesoky EA, Ebied A, Tieu T, Maraie N, Kamel MG, Ngo HT, Mattar OM, Hirayama K, Huy NT. Mast cell mediators in relation to dengue severity: A systematic review and meta-analysis. Rev Med Virol. 2020 Jan;30(1):e2084. doi: 10.1002/rmv.2084. Epub 2019 Nov 10. PMID 31709696
- [Background] Rathore AP, Mantri CK, Aman SA, Syenina A, Ooi J, Jagaraj CJ, Goh CC, Tissera H, Wilder-Smith A, Ng LG, Gubler DJ, St John AL. Dengue virus-elicited tryptase induces endothelial permeability and shock. J Clin Invest. 2019 Jul 2;129(10):4180-4193. doi: 10.1172/JCI128426. PMID 31265436
- [Background] Leo YS, Gan VC, Ng EL, Hao Y, Ng LC, Pok KY, Dimatatac F, Go CJ, Lye DC. Utility of warning signs in guiding admission and predicting severe disease in adult dengue. BMC Infect Dis. 2013 Oct 24;13:498. doi: 10.1186/1471-2334-13-498. PMID 24152678
- [Derived] Nitinai N, Nasomsong W, Chuerboonchai W, Tweekittikul A, Khingmontri V, Panuvatvanich B, Bangchuad T, Pongpraijaroen M, Roongfa-Ngarm T, Vasikasin V. Effect of montelukast in preventing dengue with warning signs among patients with dengue: A multicenter, randomized, double-blind, placebo-controlled trial. PLoS Negl Trop Dis. 2024 Feb 2;18(2):e0011927. doi: 10.1371/journal.pntd.0011927. eCollection 2024 Feb. PMID 38306389
- See also: Ahmad A, Waseem T, Butt N, Randhawa F, Malik U, Shakoori T. Montelukast Reduces the Risk of Dengue Shock Syndrome in Dengue Patients. Tropical biomedicine. 2019;35:1115-22. — https://msptm.org/files/Vol35No4/1115-1122-Tania-Shakoori.pdf